CLINICAL TRIAL: NCT06982495
Title: Comparing Two Methods for Estimating Nasogastric Tube Length: A Randomized Control Study
Brief Title: Comparing Two Methods to Measure Nasogastric Tube Length
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chiao-Hsiung Chuang, Head of Gastroenterology and Hepatology, Medical Doctor (M.D.), Doctor of Philosophy (Ph.D.), National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-BR-113-021
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Intubation, Nasogastric; Intubation Intraesophageal; Intubation Depth; Intubation Times; Intubation; Complication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCKU-NG system (Experimental): Receive nasogastric tube insertion using the NCKU-NG system (video-assisted real-time visualization, with active confirmation of passage through the esophagogastric junction and final position in the stomach based on sidehole location)
  Interventions: Device: NCKU-NG system
- Conventional blind insertion (Active Comparator): Receive traditional nasogastric tube blind bedside insertion based on standard measurement (eg. Nose-Earlobe-Xiphoid + 10 cm)
  Interventions: Other: Conventional blind insertion

INTERVENTIONS:
Device: NCKU-NG system — Nasogastric tube insertion with a novel nasogastric tube assisted placement system (NCKU-NG system)
  Arms: NCKU-NG system
Other: Conventional blind insertion — Conventional blind insertion following standard external measurement methods (eg. Nose-Earlobe-Xiphoid + 10 cm)
  Arms: Conventional blind insertion

SUMMARY:
The goal of this clinical trial is to learn if using a novel nasogastric tube assisted placement system (NCKU-NG system) can more accurately place the nasogastric tube at the optimal position in the stomach compared to conventional blind insertion techniques in adult inpatients requiring nasogastric tube placement. The main questions it aims to answer are:

* Does the NCKU-NG system improve the accuracy of nasogastric tube placement at the optimal gastric position compared to standard blind insertion?
* Does the NCKU-NG system reduce the rate of misplacement (such as entry into the airway or inadequate gastric depth), number of repeated attempts, and complication rate compared to the conventional method?
* Can estimation of nasogastric tube length using the NCKU-NG system provide a more reliable reference than external measurement or X-ray?

Researchers will compare patients randomized to nasogastric tube insertion with the NCKU-NG system (intervention arm) versus conventional blind insertion following standard external measurement methods (control arm) to see if the NCKU-NG system improves placement accuracy and reduces adverse events.

Participants will:

* Be randomized to one of two groups:

  * Intervention group: Receive nasogastric tube insertion using the NCKU-NG system (video-assisted real-time visualization, with active confirmation of passage through the esophagogastric junction and final position in the stomach based on sidehole location).
  * Control group: Receive traditional nasogastric tube blind bedside insertion based on standard measurement (eg. Nose-Earlobe-Xiphoid + 10 cm).
* All procedures will use the same material nasogastric tube (16 French polyurethane radiopaque tube).
* Undergo confirmation of tube position by X-ray within 8 hours post-insertion for both groups.
* Have the following outcomes assessed:

  * Placement accuracy (percentage of tubes placed at optimal predefined gastric position)
  * Number of placement attempts and failures
  * Rate of inadvertent airway or inadequate placement
  * Incidence of complications (e.g., aspiration, pneumothorax, gastrointestinal tract injury)
  * Correlation between video-assisted measurement and X-ray estimation of intragastric length

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥18 years)
* Patients requiring nasogastric tube placement
* Patients who are hospitalized

Exclusion Criteria:

* Patients with a chest wound that prevents palpation of the xiphoid process
* Patients who have had a gastrectomy
* Patients with a gastric tumor
* Patients with a head and neck tumor
* Patients who are agitated and difficult to place the nasogastric tube
* Patients with abnormal esophageal structure
* Patients with a basilar skull fracture
* Patients with acute upper gastrointestinal bleeding
* Patients with an expected lifespan of less than 48 hours
* Patients who cannot undergo an X-ray confirmation (e.g., pregnant women)
* Patients with unstable blood pressure (mean arterial pressure < 65 mmHg)
* Patients with ischemic, perforated, or obstructed bowel
* Patients with high-output fistula/ostomy
* Patients using photosensitive drugs
* Critically ill patients
* Patients with acute needs as determined by the attending physician
* Patients with a Glasgow Coma Scale score < 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Placement accuracy | Within 8 hours after the completion of a nasogastric tube insertion; that is, after the X-ray was taken
  Percentage of tubes placed at optimal predefined gastric position

SECONDARY OUTCOMES:
First-attempt success rate | The moment after the completion of an nasogastric tube insertion
Number of placement attempts | The moment after the completion of an nasogastric tube insertion
Insertion time | The moment after the completion of an nasogastric tube insertion
Incidence of complications | A week after the completion of an nasogastric tube insertion
Correlation between video-assisted measurement and X-ray estimation of intragastric length | Within 8 hours after the completion of an nasogastric tube insertion